CLINICAL TRIAL: NCT06379607
Title: High Flow Nasal Cannula Rates in Pediatric Asthma Exacerbations: a Feasibility Study
Brief Title: High Flow Nasal Cannula Rates in Pediatric Asthma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michele E. Smith, Assistant Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00009285
Record Dates: First submitted 2024-04-10; First posted 2024-04-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Asthma
Keywords: Asthma; High Flow Nasal Cannula; Conventional Oxygen Therapy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional Oxygen Therapy (COT) (No Intervention): Conventional Oxygen Therapy (COT) is the standard way to deliver oxygen to hypoxemic pediatric patients during an acute asthma exacerbation. Continuous albuterol will be administered via an aerogen set-up (aerogen mask, aerogen ultra, and a vibrating mesh nebulizer). Oxygen tubing will be connected to the wall and run at 2L/min as per the aerogen manufacturer's instructions.
- "Low Flow" High Flow Nasal Cannula at 4L/min (Experimental): A Fisher Paykl humidifier will be used for high flow humidification along with a flow meter and oxygen blender. A vibrating mesh nebulizer will be connected between the flow meter and the humidifier as per routine practice. Oxygen flow will be set to 4L/min and patient will be fitted with appropriately sized nasal prongs.
  Interventions: Device: "Low Flow" High Flow Nasal Cannula
- "High Flow" High Flow Nasal Cannula at 2L/kg/min (max 60L/min) (Experimental): A Fisher Paykl humidifier will be used for high flow humidification along with a flow meter and oxygen blender. A vibrating mesh nebulizer will be connected between the flow meter and the humidifier as per routine practice. Oxygen flow will be set to 2L/kg/min (max 60L/min) and patient will be fitted with appropriately sized nasal prongs.
  Interventions: Device: "High Flow" High Flow Nasal Cannula

INTERVENTIONS:
Device: "High Flow" High Flow Nasal Cannula — High Flow Nasal Cannula will be applied in both experimental groups but different flow rates will be used in each arm; this arm will use higher flow rates.
  Arms: "High Flow" High Flow Nasal Cannula at 2L/kg/min (max 60L/min)
Device: "Low Flow" High Flow Nasal Cannula — High Flow Nasal Cannula will be applied in both experimental groups but different flow rates will be used in each arm; this arm will use lower flow rates.
  Arms: "Low Flow" High Flow Nasal Cannula at 4L/min

SUMMARY:
This is a randomized, open-label, 3-armed feasibility trial will examine conventional oxygen therapy (COT) vs high flow nasal cannula at 4L/min flow vs HFNC at 2L/kg/min flow (max 60L/min) in moderate to severe pediatric asthma exacerbations.

DETAILED DESCRIPTION:
The purpose of this feasibility trial is to examine the safety and efficacy of high flow nasal cannula in moderate to severe pediatric asthma exacerbations. Eligible patients will be admitted to the Pediatric Intensive Care Unit (PICU) after initial presentation to the emergency department (ED) or as a transfer from an outside hospital ED. Patients will be admitted to the PICU on standard asthma therapy (continuous albuterol and systemic corticosteroids) based on the discretion of the treating ED physician. Upon PICU admission, eligible patients will be consented, enrolled, and randomized into the study. All patients will be continued on standard asthma therapy of continuous albuterol at 20mg/hr and systemic intravenous corticosteroids. Patient will be randomized into one of three groups: (1) conventional oxygen therapy at 2L/min via standard facemark (control group), (2) high flow nasal cannula at 4L/min, and (3) high flow nasal cannula at 2L/kg/min (max 60L/min). Pediatric Respiratory Assessment Measure (PRAM) scores and vital signs will be taken at baseline and hourly for two hours. After the two-hour long study is completed, patients will be placed on a respiratory support modality as per the treating physician's discretion. Patients will be followed longitudinally after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-17 years old with prior clinical diagnosis of asthma
* Admitted to PICU on standard asthma therapy defined as continuous albuterol and systemic corticosteroids
* Admitted to PICU on either COT or HFNC
* Admitted to PICU from either Golisano Children's Hospital ED or as a transport from an outside hospital ED within 6 hours of initial presentation
* PRAM score greater than or equal to 4 after completion of initial ED therapy

Exclusion Criteria:

* Admitted to the PICU on NIV or invasive mechanical ventilation
* Admitted to the PICU from general floors or > 6 hours from initial presentation
* Presence of a tracheostomy or baseline NIV requirement
* Pregnancy
* Immunocompromised State

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent of participants enrolled | 12 months
  Percent of participants randomized divided by the percent of participants approached.

SECONDARY OUTCOMES:
Mean Change in Pediatric Respiratory Assessment Measure (PRAM) Score | Baseline to 2 hours
  The Pediatric Respiratory Assessment Measure (PRAM) Score is a validated tool to measure asthma severity in pediatric patients. It is a scale that ranges from 0-12 with scores 4-7 indicating moderate asthma exacerbation and scores of 8-12 indicating severe exacerbation. The score has also been shown to be responsive to asthma therapies, with a decrease in score being indicative of improvement. PRAM scores will be measured at the start of the trial, at hour 1 and at the completion of the trial at hour 2. Mean changes in PRAM score will be compared across all three groups.
Mean Change in Respiratory Rate | Baseline to 2 hours
  The mean change in respiratory rate during the two our study period across all 3 study groups will be compared.
Mean Total Duration of Continuous Albuterol | Approximately 3 days
  Children will be followed longitudinally until hospital discharge and record the total duration of hours patients spent on continuous albuterol.
Percentage of Children with Escalation of Respiratory Support | 1 day
  The percentage of children requiring an increase in respiratory support (defined as escalation of support to HFNC of any flow rate, continuous positive airway pressure (CPAP), bilevel positive airway pressure (BPAP), invasive mechanical ventilation (IMV), or extracorporeal membrane oxygenation (ECMO)) either during the 2-hour trial period, immediately upon completion, or within the first 24 hours of study enrollment time will be recorded.
Mean Total Duration of Respiratory Support | Until hospital discharge, approximately 5 days
  Children will be followed longitudinally until hospital discharge and the total duration of hours patients spent on any respiratory support modality including COT, HFNC, noninvasive ventilation (NIV), invasive ventilation (IMV), or extracorporeal membrane oxygenation (ECMO) will be recorded.
Percentage of Participants placed on Adjunct Asthma Therapies | Until hospital discharge, approximately 5 days
  Investigators will describe how many children in each group were placed on adjunct asthma therapies including magnesium, heliox, leukotriene receptor antagonists, intravenous beta agonist therapies, and methylxantines either before, during, or after study period.
Percentage of Participants who needed Sedation | Until hospital discharge, approximately 5 days
  Investigators will record how many children in each group required sedation and/or anxiolytics while on their respiratory support modality either during the trial or afterwards.
Percentage of Participants on Antibiotics | Until hospital discharge, approximately 5 days
  Investigators will record how many children completed full 5-7 day courses of antibiotics for bacterial pneumonia concurrent with their asthma exacerbation.
Mean PICU Length of Stay (LOS) | Until hospital discharge, approximately 3 days
  Investigators will follow children longitudinally to record the amount of time children were admitted to the PICU for.
Mean Hospital Length of Stay (LOS) | Until hospital discharge, approximately 7 days
  Investigators will follow children longitudinally to record the amount of time children were admitted to the hospital for.

CONTACTS AND LOCATIONS:
Overall Officials: MicheleE E Smith, MD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of Rochester Golisano Children's Hospital, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No